CLINICAL TRIAL: NCT02218320
Title: A Phase IV, Open-Label Study to Compare Virologic and Immunologic Responses to Raltegravir and Dolutegravir in the Gastrointestinal Tract of HIV-Positive Men and Women
Brief Title: Comparison of Virologic and Immunologic Responses to Raltegravir and Dolutegravir in the Gastrointestinal Tract of HIV-Positive Adults
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-1647
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2017-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Gut-associated lymphoid tissue; raltegravir; Isentress; dolutegravir; Tivicay; pharmacodynamics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; dolutegravir; Colonoscopy; Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Ten HIV-infected adults will be in Group A and take the HIV medication raltegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Interventions: Drug: Raltegravir; Procedure: Colonoscopy with biopsy
- Group B: Ten HIV-infected adults will be in Group B and take the HIV medication dolutegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Interventions: Drug: Dolutegravir; Procedure: Colonoscopy with biopsy

INTERVENTIONS:
Drug: Raltegravir
  Other Names: Isentress ®
  Groups: Group A
Drug: Dolutegravir
  Other Names: Tivicay ®
  Groups: Group B
Procedure: Colonoscopy with biopsy — This procedure is not standard of care for patients receiving combination antiretroviral therapy (cART), but is necessary to obtain tissue samples.

SUMMARY:
This is a Phase IV, open label, observational study to compare the gastrointestinal tissue concentrations, inflammatory response, and viral replication of two integrase-inhibitors, raltegravir and dolutegravir, in HIV-infected volunteers who are virologically suppressed in blood plasma. The study will be comprised of 20 HIV-infected volunteers who will be enrolled equally into two groups. Group A will consist of 10 subjects receiving an antiretroviral regimen of tenofovir, emtricitabine, and raltegravir, and Group B will consist of 10 subjects receiving an antiretroviral regimen of tenofovir, emtricitabine, and dolutegravir. Participants will provide small pieces of tissue, or biopsies, which will be taken from three distinct locations of the large intestine during a colonoscopy procedure. These biopsies will be used to measure the amount of raltegravir or dolutegravir, HIV virus, and inflammatory markers present in the gastrointestinal tract.

DETAILED DESCRIPTION:
Purpose: To compare virologic and immunologic responses to raltegravir and dolutegravir in the gastrointestinal tract of HIV-positive men and women

Participants: Twenty HIV-infected volunteers will be enrolled equally into two groups. Group A will consist of subjects receiving an antiretroviral regimen of raltegravir, tenofovir, and emtricitabine and Group B will consist of subjects receiving an antiretroviral regimen of dolutegravir, tenofovir, and emtricitabine.

Procedures (methods): This is a Phase IV, open label study to compare the gastrointestinal tissue concentrations, cytokine response, and viral replication in gut-associated lymphoid tissue of two integrase-inhibitors in HIV-infected volunteers who are virologically suppressed in blood plasma. Subjects will undergo an observed bowel preparation, followed by a colonoscopy in which tissue will be obtained by a board-certified gastroenterologist from the terminal ileum/ascending colon, splenic flexture, and rectum/sigmoid colon. Blood plasma will be collected immediately prior to collection of tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy HIV-positive adults aged 18-65, inclusive on the date of screening, with documentation of at least one positive HIV test. Healthy is defined as no clinically relevant abnormalities that would interfere with the interpretation of results, or pose unnecessary risk onto volunteers due to study procedures.
* Receiving an antiretroviral regimen containing tenofovir+emtricitabine with raltegravir (Group A) or dolutegravir (Group B) for > 3 months, with blood plasma HIV RNA < 50copies/mL for at least 4 weeks, or a 2 log decrease in baseline blood plasma HIV RNA.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Documentation of at least 80% adherence to antiretroviral regimen, through clinician or self-report, with no missed doses in the 3 days prior to the inpatient visit.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
* Women of childbearing potential must be utilizing at least one acceptable form of birth control.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurologic disease that would pose unnecessary risk or interfere with study results. Subjects will be excluded for any condition that would increase risk from sedation, endoscopy, or biopsy.
* Subjects with a history of having a gastrectomy, colostomy, ileostomy, or any other clinically significant procedure altering the gastrointestinal tract, or any condition possibly affecting drug absorption.
* Subjects with inflammatory bowel diseases (ulcerative colitis or Crohn's disease).
* Female subjects who are currently pregnant or breastfeeding, or planning to become pregnant during the study period.
* Subjects who are unwilling to refrain from insertion of medical/recreation devices and products into the rectum, and from receptive anal intercourse, for 72 hours before inpatient study visit and through 7 days after the last biopsy unless instructed otherwise by the investigators.
* A positive urine drug screen.
* Untreated rectal sexually transmitted infection at screening.
* Treatment with an investigational drug within 2 months preceding study enrollment.
* Participated in a gastrointestinal biopsy study in the 3 months preceding study enrollment.
* Participants with a history of clotting or bleeding disorders.
* Participants with a history of abnormal reaction to, or complication from, conscious sedation or anesthesia
* Subjects who are unwilling or unable to comply with the following dietary restrictions in regard to study procedures, including a clear liquid diet during bowel preparation and a period of NPO (nil per os) prior to the colonoscopy. While confined, the total daily nutritional composition will be 50% carbohydrate, 15% protein, and 35% fat. The daily caloric intake should not exceed 3200kcal.
* Abnormalities of the colorectal mucosa, or significant colorectal symptom(s), which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids).
* Any other reason or condition that in the judgment of the investigators would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from University of North Carolina Infectious Diseases Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Clinical and Translational Research Center, UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weber MD, Andrews E, Prince HA, Sykes C, Rosen EP, Bay C, Shaheen NJ, Madanick RD, Dellon ES, De Paris K, Nelson JA, Gay CL, Kashuba AD. Virological and immunological responses to raltegravir and dolutegravir in the gut-associated lymphoid tissue of HIV-infected men and women. Antivir Ther. 2018;23(6):495-504. doi: 10.3851/IMP3236. PMID 29714167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began upon IRB approval. Patients were enrolled from December 2014 to October 2015, at which time data analysis ensued. Enrollment continued until 20 subjects completed all study procedures. Patients were recruited from the Infectious Disease clinics associated with the University of North Carolina at Chapel Hill.
Pre-assignment Details: After informed consent, all patients underwent a screening visit to determine eligibility. This visit had to occur within the 6 weeks prior to study enrollment. Patients were enrolled into the group that matched their treatment regimen.
Groups:
- Group A: Ten HIV-infected adults will be in Group A and take the HIV medication raltegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Raltegravir
  Colonoscopy with biopsy: This procedure is not standard of care for patients receiving combination antiretroviral therapy (cART), but is necessary to obtain tissue samples.
- Group B: Ten HIV-infected adults will be in Group B and take the HIV medication dolutegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Dolutegravir
  Colonoscopy with biopsy: This procedure is not standard of care for patients receiving combination antiretroviral therapy (cART), but is necessary to obtain tissue samples.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 10 (First participant visit on this arm Dec 2014) | 10 (First participant contact on this arm was December 2014)
Completed | 10 (Last participant contact on this arm was June 2015) | 10 (Last participant contact on this arm was October 2015)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Ten HIV-infected adults will be in Group A and take the HIV medication raltegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Raltegravir
  Colonoscopy with biopsy: This procedure is not standard of care for patients receiving combination antiretroviral therapy (cART), but is necessary to obtain tissue samples. All 10 subjects underwent a bowel prep with subsequent colonoscopy to obtain tissue samples.
- Group B: Ten HIV-infected adults will be in Group B and take the HIV medication dolutegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Dolutegravir
  Colonoscopy with biopsy: This procedure is not standard of care for patients receiving combination antiretroviral therapy (cART), but is necessary to obtain tissue samples. All 10 subjects underwent a bowel prep with subsequent colonoscopy to obtain tissue samples.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 54.5 [48 to 64] | 49.5 [32 to 56] | 52.5 [32 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 3 | 3 | 6
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Rectal Tissue Concentrations of Ralegravir and Dolutegravir
Time Frame: 2 to 6 hours post dose
Measure: Median (Full Range); unit: ng/g
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
ng/g | 5308 [3938 to 19600] | 810 [510 to 1408]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney)

2. Primary Outcome: RNA Concentrations From Gastrointestinal Tissues
Description: We measured RNA concentrations in copies/1000cells for both drug groups
Time Frame: 2 to 6 hours post dose
Measure: Median (Full Range); unit: copies/1000cells
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
copies/1000cells | 0.05 [0.03 to 0.34] | 0.16 [0.01 to 36.19]

3. Primary Outcome: Percentage of Total CD8+ T-cells With CCR5 Expression
Description: Local immunologic markers in gastrointestinal tract tissues
Time Frame: 2 to 6 hours post dose
Measure: Median (Full Range); unit: percentage of total cells
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
percentage of total cells | 0.15 [0.07 to 0.52] | 0.64 [0.24 to 1.60]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent at the screening visit (up to 42 days prior to enrollment) through study completion (Up to 14 days after last sampling).
Description: Adverse events were assessed at all visits with a standardized IRB-approved questionnaire.
Groups:
- Group A: Ten HIV-infected adults will be in Group A and take the HIV medication raltegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Raltegravir
  Colonoscopy with biopsy: This procedure is not standard of care for patients receiving combination antiretroviral therapy (cART), but is necessary to obtain tissue samples. All participants underwent a bowel prep with subsequent colonoscopy to obtain tissue samples.
- Group B: Ten HIV-infected adults will be in Group B and take the HIV medication dolutegravir in combination with tenofovir and emtricitabine as their provider-prescribed antiretroviral regimen.
  Dolutegravir
  Colonoscopy with biopsy: This procedure is not standard of care for patients receiving combination antiretroviral therapy (cART), but is necessary to obtain tissue samples.All participants underwent a bowel prep with subsequent colonoscopy to obtain tissue samples.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=10) | Group B (N=10)
Thombophlebitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Onset 26Apr15, resolution 15May15, treated with Clindamycin
Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Elevated reading of blood pressure were noted on study, beginning 04May2015. Participant referred to PCP for management.
Anal Irritation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Onset and resolution 28Jan2015. Participant used aloe wipe on anus and symptoms resolved.
Abdominal gas cramps (Gastrointestinal disorders) | 1 (1) | 1 (1) — Onset and resolution 06Jan2015. Patient ambulated to resolution of symptoms with one dose of Tylenol.
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Onset 13Dec14 and resolution 18Dec14. Resolved without treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No